CLINICAL TRIAL: NCT04231877
Title: A Pilot Study to Estimate the Safety and Tolerability of the Combination of Polatuzumab Vedotin, With or Without Glofitamab, With Dose Adjusted Rituximab, Etoposide, Cyclophosphamide, and Doxorubicin (PERCH) for Upfront Treatment of Aggressive B-Cell Non-Hodgkin Lymphomas
Brief Title: Polatuzumab Vedotin and Combination Chemotherapy With or Without Glofitamab for the Treatment of Untreated Aggressive Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1006477; NCI-2019-08983 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10423 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; ALK-Positive Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Primary Mediastinal Large B-Cell Lymphoma; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Gray-Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Prednisone; deltacortene; Etoposide; Doxorubicin; Cyclophosphamide; glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (polatuzumab vedotin, chemotherapy) [CLOSED TO ACCRUAL 05/23/2024] (Experimental): Patients receive rituximab IV on day 1, polatuzumab vedotin IV on day 1, prednisone PO BID on days 1-5, etoposide IV on days 1-4, doxorubicin IV on days 1-4, and cyclophosphamide IV on day 5. Patients also receive filgrastim SC 24-72 hours after the last dose of each treatment cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo MUGA scan or echocardiography during screening and FDG PET, CT scan, bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Drug: Polatuzumab Vedotin; Biological: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography; Procedure: FDG-Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration
- Arm B (polatuzumab vedotin, glofitamab, chemotherapy) (Experimental): Patients receive rituximab IV on day 1, polatuzumab vedotin IV on day 1, prednisone PO BID on days 1-5, etoposide IV on days 1-4, doxorubicin IV on days 1-4, and cyclophosphamide IV on day 5. Starting with cycle 2, patients also receive glofitamab, over 4 hours, on day 1 and 8 of cycle 2 and day 1 of subsequent cycles. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo MUGA scan or echocardiography during screening and FDG PET, CT scan, bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Drug: Polatuzumab Vedotin; Biological: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Biological: Glofitamab; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography; Procedure: FDG-Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Given IV
  Other Names: 1313206-42-6; ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
Biological: Rituximab — Given IV
  Other Names: 174722-31-7; 687451; ABP 798; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-C2B8 Monoclonal Antibody; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; rituximab-abbs; Rituximab Biosimilar SIBP-02; Riabni; Rituximab ARRX; Rituximab PVVR; Ruxience
Drug: Prednisone — Given PO
  Other Names: 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Metacortandracin; Meticorten; Ofisolona; Panafcort; Paracort; Predicor; Predicorten; Prednidib; Prednilonga; Prednitone
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin
Biological: Glofitamab — Given IV
  Other Names: Glofitamab-gxbm; RO7082859
  Arms: Arm B (polatuzumab vedotin, glofitamab, chemotherapy)
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: MUGA Scan; MUGA
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET scan
  Other Names: FDG-PET; FDG-PET Imaging
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT Scan; CT Scan; Computed Axial Tomography
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration

SUMMARY:
This phase I trial studies the side effects of polatuzumab vedotin when given with combination chemotherapy with or without glofitamab for the treatment of patients with untreated large B-cell lymphoma that grows and spreads quickly and has severe symptoms (aggressive). Polatuzumab vedotin is a monoclonal antibody, polatuzumab, linked to a toxic agent called vedotin. Polatuzumab attaches to CD79B positive cancer cells in a targeted way and delivers vedotin to kill them. Glofitamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Drugs used in combination chemotherapy such as etoposide, cyclophosphamide, and doxorubicin work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Anti-inflammatory drugs, such as prednisone, lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving polatuzumab vedotin in combination chemotherapy with or without glofitamab may help treat patients with aggressive large B-cell lymphoma.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A (CLOSED TO ACCRUAL 05/23/2024): Patients receive rituximab intravenously (IV) on day 1, polatuzumab vedotin IV on day 1, prednisone orally (PO) twice daily (BID) on days 1-5, etoposide IV on days 1-4, doxorubicin IV on days 1-4, and cyclophosphamide IV on day 5. Patients also receive filgrastim subcutaneously (SC) 24-72 hours after the last dose of each treatment cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo multigated acquisition (MUGA) scan or echocardiography during screening and fludeoxyglucose (FDG) positron emission tomography (PET), computed tomography (CT) scan, bone marrow biopsy and aspiration and blood sample collection throughout the study.

ARM B: Patients receive rituximab IV on day 1, polatuzumab vedotin IV on day 1, prednisone PO BID on days 1-5, etoposide IV on days 1-4, doxorubicin IV on days 1-4, and cyclophosphamide IV on day 5. Starting with cycle 2, patients also receive glofitamab, over 4 hours, on day 1 and 8 of cycle 2 and day 1 of subsequent cycles. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MUGA scan or echocardiography during screening and FDG PET, CT scan, bone marrow biopsy and aspiration and blood sample collection throughout the study.

After the completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Untreated aggressive B-cell large-B cell lymphoma (non-Hodgkin lymphoma) with adverse features that may predict sub-optimal response to rituximab-cyclophosphamide, doxorubicin (hydroxydaunorubicin), vincristine (Oncovin), prednisone (R-CHOP) and in the opinion of the investigator would be treated with DA-EPOCH-R as standard of care. Subjects must be planned to receive full course (6 cycles) chemoimmunotherapy as per clinical standard of care. Composite lymphomas are not excluded provided that the subject has not receive prior systemic therapy for the indolent component and would receive DA-EPOCH-R as the standard of care regimen for the aggressive component. Eligible histologies based on 2016 World Health Organization (WHO) classification include:

  * High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 translocations
  * High grade B-cell lymphoma, not otherwise specified (NOS)
  * Diffuse large B-cell lymphoma (DLBCL) NOS
  * Primary mediastinal B-cell lymphoma
  * T-cell/histiocyte-rich large-B-cell lymphoma
  * Epstein-Barr virus (EBV) + DLBCL, NOS
  * ALK+ large B-cell lymphoma (must be CD20+)
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
* Be willing and able to provide written informed consent for the trial
* Be >= 18 years of age on day of signing informed consent
* Have measurable disease, including at least 1 nodal site measuring 1.5 cm or 1 extranodal site measuring 1.0 cm in longest dimension on computed tomography (CT) or fluorodeoxyglucose-positron emission tomography (FDG-PET)
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale (PS)
* Left ventricular ejection fraction (LVEF) >= 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Absolute neutrophil count (ANC) >= 1,000/uL except in cases of marrow infiltration by lymphoma
* Platelets >= 75,000 / mcL except in cases of marrow infiltration by lymphoma or hypersplenism
* Hemoglobin >= 8 g/dL except in cases of marrow infiltration by lymphoma without red blood cell (RBC) transfusion within 14 days of first treatment
* Measured or calculated creatinine clearance (Glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 40 mL/min.

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN) (Patients with documented Gilbert disease may be enrolled if total bilirubin =< 3.0 x ULN)
* Direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver involvement
* International Normalized Ratio (INR) or Prothrombin Time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants, or subject is shown to have an antiphospholipid antibody on workup
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of =< 1% per year during the treatment period and for at least 12 months after the last dose of EPCH-R, 9 months after the last dose of polatuzumab, 2 months after the last dose of glofitamab (Arm B participants), or 3 months after the last dose of tocilizumab (if applicable), whichever is longer. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (=<12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements. Examples of contraceptive methods with a failure rate of =<1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
* For women of childbearing potential, a negative serum pregnancy test result during screening period. Women who are considered not to be of childbearing potential are not required to have a pregnancy test
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of EPCH-R or polatuzumab, 2 months after the last dose of glofitamab (Arm B participants), or 2 months after the last dose of tocilizumab (if applicable), whichever is longer. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. Male patients considering preservation of fertility should bank sperm before study treatment
* ARM B ONLY: Negative SARS-CoV-2 antigen or PCR test within 7 days prior to enrollment

Exclusion Criteria:

* Contraindication to any of the individual components of glofitamab, tocilizumab or EPCH-R, including prior receipt of anthracyclines, or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, or known sensitivity or allergy to murine products
* Prior systemic treatment for lymphoma with the exception of corticosteroids. Prior radiotherapy is allowed provided that this site is not used as a measurable site to assess response.
* Richter's transformation from chronic lymphocytic leukemia/small lymphocytic lymphoma is not allowed. Transformation from follicular or other indolent lymphomas is allowed provided that the subject has not received prior systemic therapy for their lymphoma and the aggressive component meets one of the criteria listed in inclusion criterion 1
* Diagnosis of Burkitt lymphoma
* Prior organ transplantation
* Current Grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
* Prior systemic therapy for indolent lymphoma
* Prior use of any monoclonal antibody within 3 months of the start of cycle 1; any investigational therapy within 28 days prior to the start of cycle 1; vaccination with live vaccines within 28 days prior the start of cycle 1 and at any time during the study treatment period
* Prior therapy for large B-cell lymphoma except for patients who require lymphoma symptom control during screening may receive steroids in the following manner: Up to 30 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening, including prior to finalization of staging (not included as part of pre-phase treatment) If glucocorticoid treatment is urgently required at higher doses for lymphoma symptom control prior to the start of study treatment, tumor assessments must be completed prior to initiation of > 30-100 mg/day of prednisone or equivalent. Prednisone > 30-100 mg/day or equivalent may be given for a maximum of 7 days as a pre-phase treatment. If patients exceed the allowed dosing of corticosteroids, patients may still be eligible for the study provided that baseline imaging is performed (or repeated) after completion of the course of higher dose of steroids. Allowed corticosteroid dosing resets from the point of imaging forward and patients who do not exceed the allowed corticosteroid dosing from the point of imaging until initiation of study treatment may enroll
* History of other malignancy that could affect compliance with the protocol or interpretation of results except with permission of the principal investigator. The following are eligible without a specific waiver:

  * Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible
  * Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for >= 2 years prior to enrollment are eligible
  * Patients with low-grade, early-stage prostate cancer (Gleason score 6 or below, Stage 1 or 2) with no requirement for therapy at any time prior to study are eligible
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Recent major surgery (within 4 weeks prior to the start of cycle 1), other than for diagnosis
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) which requires systemic treatment. Patients may proceed with screening during treatment for infection, but systemic treatment must be completed by cycle 1 day 1
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology):

  * Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) DNA is undetectable at the time of screening. These patients must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated by institutional standard
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)

  * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History of uncontrolled human immunodeficiency virus (HIV)

  * Patients with known diagnosis of HIV must have undetectable viral load, have a CD4 count ≥ 200/μL, and be on anti-retroviral therapy. HIV positive patients should be monitored per local/institutional standards while receiving study treatment
* Patients with a history of progressive multifocal leukoencephalopathy
* Pregnancy or lactation or intending to become pregnant during study
* ARM B ONLY: Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* ARM B ONLY: Known or suspected chronic active Epstein-Barr virus infection
* ARM B ONLY: Current or past history of Waldenström macroglobulinemia
* ARM B ONLY: Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, CNS lymphoma or neurodegenerative disease
* ARM B ONLY: Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurological deficits, as judged by the investigator, are allowed
* ARM B ONLY: Active autoimmune disease which is not well controlled by therapy
* ARM B ONLY: Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible
* ARM B ONLY: Participants with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
* ARM B ONLY: Participants with active autoimmune disease with dermatologic manifestations are eligible for the study
* ARM B ONLY: Participants with a history of autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, multiple sclerosis, or glomerulonephritis will be excluded
* ARM B ONLY: Participants with a history of immune thrombocytopenic purpura, autoimmune hemolytic anemia, Guillain-Barré syndrome, myasthenia gravis, myositis, rheumatoid arthritis, vasculitis, or other autoimmune disease will be excluded unless they have not required systemic therapy in the last 12 months
* ARM B ONLY: Clinically significant liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* ARM B ONLY: Suspected active or latent tuberculosis (as confirmed by a positive interferon-gamma release assay)
* ARM B ONLY: Grade 3 infection within 4 weeks of treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of polatuzumab or first administration of alternate therapy
  Will estimate the safety and tolerability of polatuzumab vedotin when added to dose-adjusted-etoposide, prednisone, vincristine (Oncovin), cyclophosphamide, doxorubicin-rituximab (DA-EPCH-R) with or without glofitamab, chemoimmunotherapy.

SECONDARY OUTCOMES:
The proportion of patients who are unable to complete 6 cycles of therapy for reasons other than disease progression | Up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lynch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roschewski M, Kurtz DM, Westin JR, Lynch RC, Gopal AK, Alig SK, Sworder BJ, Cherng HJ, Kuffer C, Blair D, Brown K, Goldstein JS, Schultz A, Close S, Chabon JJ, Diehn M, Wilson WH, Alizadeh AA. Remission Assessment by Circulating Tumor DNA in Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec;43(34):3652-3661. doi: 10.1200/JCO-25-01534. Epub 2025 Aug 13. PMID 40802906
- [Derived] Lynch RC, Poh C, Ujjani CS, Warren EH, Smith SD, Shadman M, Morris K, Lee S, Rasmussen H, Ottemiller S, Shelby M, Keo S, Verni K, Kurtz DM, Alizadeh AA, Chabon JJ, Hogan GJ, Schulz A, Gooley T, Voutsinas JM, Gopal AK. Polatuzumab vedotin with infusional chemotherapy for untreated aggressive B-cell non-Hodgkin lymphomas. Blood Adv. 2023 Jun 13;7(11):2449-2458. doi: 10.1182/bloodadvances.2022009145. PMID 36521030